CLINICAL TRIAL: NCT00301860
Title: Feasibility of Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation Followed by Donor Lymphocyte Infusions for Children at High Risk for Complications With Conventional Transplantation
Brief Title: Donor Stem Cell Transplant Followed By Donor White Blood Cell Infusions in Treating Young Patients With Hematologic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462439; UCSF-02164; UCSF-H10216-21819-03
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma
Keywords: childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood small noncleaved cell lymphoma; juvenile myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Dendritic Cell Sarcoma, Interdigitating; Recurrence | interventions — Antilymphocyte Serum; Filgrastim; Cyclosporine; fludarabine phosphate; Melphalan; Methotrexate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Drug: methotrexate
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor peripheral blood stem cell transplant helps stop both the growth of cancer cells and the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving chemotherapy, such as fludarabine and melphalan, and antithymocyte globulin before transplant and cyclosporine and methotrexate after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well donor stem cell transplant, using low-dose chemotherapy and antithymocyte globulin, followed by donor white blood cell infusions work in treating young patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of allogeneic hematopoietic stem cell transplantation using a reduced-intensity conditioning regimen, in terms of whole blood engraftment rate at 100 days post transplant, in pediatric patients with hematopoietic malignancies who are at high risk for complications with conventional transplantation.
* Determine the feasibility of donor lymphocyte infusions (DLIs), in terms of number of patients who receive at least one DLI by 12 months post transplant, in patients treated with this regimen.
* Determine the toxicities of the conditioning regimen, in terms of 100-day post transplant nonrelapse-related death rate, in these patients.
* Determine the toxicity of DLI, in terms of acute and chronic graft-vs-host disease rate and 12-month post transplant nonrelapse-related death rate, in these patients.

OUTLINE: This is a pilot study.

* Reduced-intensity conditioning regimen: Patients receive fludarabine IV on days -6 to -2; antithymocyte globulin IV on days -5 to -2; and melphalan IV on days -3 and -2.
* Transplantation: Patients undergo allogeneic peripheral blood stem cell transplantation on day 0. Patients also receive filgrastim (G-CSF) IV beginning on day 5 and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV or orally beginning on day -1 and continuing until at least day 28 and methotrexate IV on days 1, 3, and 6.
* Donor lymphocyte infusion (DLI): Patients with mixed chimerism, no acute GVHD requiring therapy, and no relapse/progression post transplant at day 90 may receive DLI. At least 30 days after discontinuation of immunosuppression, patients may receive up to 2 DLIs at least 8-12 weeks apart in the absence of GVHD.

At the completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematopoietic malignancies:

  * Acute lymphoblastic leukemia or myeloid leukemia with < 30% blasts in the bone marrow
  * Juvenile myelomonocytic leukemia
  * Chronic myelogenous leukemia in chronic or accelerated phase
  * Relapsed non-Hodgkin's or Hodgkin's lymphoma in at least partial remission
* Considered at high risk (> 30%) of toxic death with standard hematopoietic stem cell transplantation (HSCT), as indicated by at least one of the following:

  * Creatinine > 1.5 times normal OR creatinine clearance < 70 mL/min OR tubular damage that is not corrected by cessation of chemotherapy
  * DLCO < 60% of predicted OR history of prior intubation due to lung disease (intubation for surgery excluded)
  * Shortening fraction < 30%
  * History of disseminated fungal infection during chemotherapy OR currently receiving antifungal agents OR history of ≥ 2 septic episodes (confirmed by cultures) that required ICU support

    * Patients with improving fungal or other infections eligible

      * Improving infection is defined as confirmed negative cultures on 2 separate occasions, at least 1 week apart, and/or stable or improving imaging studies (e.g., CT scan) of the infected site
      * Two imaging studies taken at least 2 weeks apart must show stable or improved disease
  * History of stroke or abnormal MRI/MRA OR leukoencephalopathy OR seizures that are not fully controlled with anticonvulsants (> 2 episodes of seizures in the preceding year or 1 episode of status epilepticus in a patient who is receiving anticonvulsant therapy)
  * History of prior significant bleeding (e.g., pulmonary, CNS, or gastrointestinal) OR history of a clotting disorder as manifested by prior significant thromboses (e.g., superior vena cava, inferior vena cava, or femoral vein)
* Failed conventional therapies and not eligible for myeloablative protocols

  * May have failed prior conventional HSCT
* No active CNS leukemia
* Unrelated or related donor available, meeting the following criteria:

  * Matched for at least 7/8 loci by high-resolution typing
  * One mismatch at A, B, or C loci allowed
  * Fully matched at DRB1 locus

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* No active/progressing viral, bacterial, protozoal, or fungal infection
* Transaminases ≤ 5 times normal (except in the presence of autoimmune liver disease)
* Shortening fraction ≥ 25%
* DLCO ≥ 40% OR pulse oximetry ≥ 85% on room air
* Glomerular filtration rate ≥ 40 mL/min

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior prolonged intensive chemotherapy (> 3 years of therapy or ≥ 3 different chemotherapeutic protocols) allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2003-01; Primary Completion 2007-03 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Horn, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States